CLINICAL TRIAL: NCT07168577
Title: Evaluation of Sleep Quality and Caregiver Burden in Children With Cerebral Palsy
Brief Title: Sleep Quality and Caregiver Burden in Children With Cerebral Palsy
Acronym: CP-SLEEP
Status: Not yet recruiting | Type: Observational
Sponsor: Selim Sezikli (Other Government)
Responsible Party: Sponsor-Investigator, Selim Sezikli, Medical Doctor, Specialist in Physical Medicine and Rehabilitation, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Organization: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Other Study IDs: CP-2025-01
Record Dates: First submitted 2025-09-05; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Cerebral Palsy; Sleep Disorders in Children; Caregiver Burden; Sleep Quality; Anxiety and Depression (Caregivers)
Keywords: Zarit Burden Interview (ZBI); Children's Sleep Habits Questionnaire (CSHQ); Cerebral palsy; Sleep quality; Pittsburgh Sleep Quality Index (PSQI); Sleep disorders; Caregiver burden; Caregiver sleep quality
MeSH Terms: conditions — Cerebral Palsy; Caregiver Burden; Sleep Initiation and Maintenance Disorders; Anxiety Disorders; Depression; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children With Cerebral Palsy and Primary Caregivers: This cohort includes children aged 2-18 years with a confirmed diagnosis of cerebral palsy and their primary caregivers (parents or legal guardians aged ≥18 years). All participants will undergo standardized clinical and questionnaire-based assessments. For children, sleep quality will be evaluated with the Children's Sleep Habits Questionnaire (CSHQ), and functional status will be classified using GMFCS, MACS, and CFCS, while spasticity will be assessed with the Modified Ashworth Scale. For caregivers, sleep quality will be assessed with the Pittsburgh Sleep Quality Index (PSQI), caregiver burden with the Zarit Burden Interview (ZBI), and psychological status with the Hospital Anxiety and Depression Scale (HADS). No experimental intervention will be applied; the study is observational and cross-sectional.

SUMMARY:
Cerebral palsy (CP) is a lifelong condition that affects movement and posture in children, often requiring continuous care from family members. Children with CP frequently experience sleep problems due to spasticity, pain, seizures, or behavioral difficulties. Poor sleep can negatively affect the child's health and development, as well as increase the physical and emotional burden on their caregivers.

This study aims to evaluate the sleep quality of children with CP and their primary caregivers, and to examine the relationship between caregiver burden and these sleep-related factors. The study will include children aged 2 to 18 years with a diagnosis of CP and their primary caregivers (parents or legal guardians).

Children's sleep patterns will be assessed using the Children's Sleep Habits Questionnaire (CSHQ). Their functional levels will be classified using the Gross Motor Function Classification System (GMFCS), Manual Ability Classification System (MACS), and Communication Function Classification System (CFCS). Caregivers' sleep quality will be assessed with the Pittsburgh Sleep Quality Index (PSQI), caregiver burden with the Zarit Burden Interview (ZBI), and psychological status with the Hospital Anxiety and Depression Scale (HADS).

By identifying how sleep problems are linked with caregiver burden and psychological health, this study may provide valuable insights for developing supportive intervention programs for both children with CP and their families.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is the most common cause of motor disability in childhood and often requires long-term daily care provided by family members. Sleep disorders are highly prevalent in children with CP compared with typically developing peers and are frequently associated with spasticity, seizures, pain, and behavioral issues. Poor sleep may further compromise the child's functional capacity and quality of life. At the same time, caregivers of children with CP often face increased physical and psychological demands, including high levels of stress, anxiety, and depression, which may be exacerbated by poor sleep quality and increased caregiving burden.

Although prior studies have investigated these factors separately, there is limited research examining the combined relationship between child sleep quality, functional status, caregiver sleep quality, caregiver burden, and psychological health. A comprehensive evaluation of these interrelated aspects may help in identifying high-risk groups and developing supportive interventions for both children and caregivers.

This single-center, observational, cross-sectional study will be conducted in the outpatient Physical Medicine and Rehabilitation clinics of Istanbul Physical Medicine and Rehabilitation Training and Research Hospital. The study will recruit at least 100 child-caregiver pairs. Children aged 2-18 years with a confirmed diagnosis of CP and their primary caregivers (aged ≥18 years) will be included. Sampling will be based on convenience and voluntary participation.

Data collection will include standardized questionnaires and clinical classifications. For children, sleep quality will be assessed using the Children's Sleep Habits Questionnaire (CSHQ), while functional levels will be determined by the Gross Motor Function Classification System (GMFCS), Manual Ability Classification System (MACS), and Communication Function Classification System (CFCS). Spasticity will be evaluated with the Modified Ashworth Scale. For caregivers, sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI), caregiver burden with the Zarit Burden Interview (ZBI), and psychological status with the Hospital Anxiety and Depression Scale (HADS).

All assessments will be performed by trained researchers through face-to-face interviews following standardized protocols. Data will be analyzed using descriptive statistics, correlation tests, and multivariable regression analyses to explore the associations between child sleep quality, caregiver sleep quality, caregiver burden, and psychological outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2-18 years with a confirmed diagnosis of cerebral palsy
* Primary caregiver (≥18 years, parent or legal guardian) responsible for the child's daily care
* Ability to read and write in Turkish
* Sufficient cognitive capacity to complete questionnaires and participate in interviews
* Voluntary agreement of both the child's caregiver and participant to join the study

Exclusion Criteria:

* Presence of severe comorbid neurological or metabolic disease in the child
* Caregiver with a history of severe psychiatric disorder or cognitive impairment
* Communication problems that prevent completion of questionnaires
* Hospitalization within the last 3 months due to acute medical condition
* Withdrawal of consent or incomplete questionnaires during the study

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of children aged 2-18 years diagnosed with cerebral palsy and their primary caregivers (parents or legal guardians aged ≥18 years). Participants will be recruited from the outpatient clinics of Istanbul Physical Medicine and Rehabilitation Training and Research Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-09-08 (Estimated); Primary Completion 2026-03-08 (Estimated); Study Completion 2026-03-08 (Estimated)

PRIMARY OUTCOMES:
Child Sleep Quality Assessed by Children's Sleep Habits Questionnaire (CSHQ) | Day 1 (single assessment at baseline)
  Sleep quality of children with cerebral palsy will be assessed using the parent-reported Children's Sleep Habits Questionnaire (CSHQ), a validated scale measuring common sleep behaviors and problems in children.
Caregiver Sleep Quality Assessed by Pittsburgh Sleep Quality Index (PSQI) | Day 1 (single assessment at baseline)
  Sleep quality of caregivers will be measured using the Pittsburgh Sleep Quality Index (PSQI), which evaluates sleep patterns and disturbances over the previous month.
Caregiver Burden Assessed by Zarit Burden Interview (ZBI) | Day 1 (single assessment at baseline)
  Caregiver burden will be assessed using the Zarit Burden Interview (ZBI), a validated questionnaire evaluating the impact of caregiving on emotional, physical, and social well-being.

SECONDARY OUTCOMES:
Child Functional Level Assessed by Gross Motor Function Classification System (GMFCS) | Day 1 (single assessment at baseline)
  Functional motor levels of children with cerebral palsy will be classified according to the GMFCS, a standardized 5-level system describing gross motor function.
Manual Ability Assessed by Manual Ability Classification System (MACS) | Day 1 (single assessment at baseline)
  Hand function and manual ability of children will be evaluated using the MACS, a validated classification system for children with cerebral palsy.
Communication Function Assessed by Communication Function Classification System (CFCS) | Day 1 (single assessment at baseline)
  Communication ability of children will be assessed using the CFCS, which categorizes functional communication performance in daily life.
Spasticity Assessed by Modified Ashworth Scale (MAS) | Day 1 (single assessment at baseline)
  Muscle spasticity will be measured using the Modified Ashworth Scale (MAS), a widely used clinical tool for grading resistance to passive movement.
Caregiver Psychological Status Assessed by Hospital Anxiety and Depression Scale (HADS) | Day 1 (single assessment at baseline)
  Caregivers' psychological health will be evaluated using the HADS, a self-reported screening tool for symptoms of anxiety and depression.

CONTACTS AND LOCATIONS:
Overall Officials: Selim Sezikli, MD, Principal Investigator — Istanbul Physical Medicine and Rehabilitation Training and Research Hospital
Locations (1):
- Istanbul Physical Medicine and Rehabilitation Training and research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared, including demographic information, child sleep quality scores (CSHQ), functional classification levels (GMFCS, MACS, CFCS), spasticity scores (MAS), caregiver sleep quality (PSQI), caregiver burden (ZBI), and psychological status (HADS). Data will be anonymized and shared in compliance with ethical and confidentiality requirements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified individual participant data and supporting documents (study protocol, SAP, ICF) will be available beginning 6 months after study completion (September 2026) and will remain available for 2 years (until March 2028).
Access Criteria: Qualified researchers who have obtained approval from an independent ethics committee and signed a data use agreement will be able to access the de-identified individual participant data (IPD) and supporting information (study protocol, statistical analysis plan, informed consent form). Data will include demographic characteristics, child sleep quality (CSHQ), functional classification (GMFCS, MACS, CFCS), spasticity (MAS), caregiver sleep quality (PSQI), caregiver burden (ZBI), and psychological status (HADS). All data will be provided in anonymized form to protect confidentiality. Access requests should be submitted to the principal investigator, and approved researchers will receive data electronically.